CLINICAL TRIAL: NCT02060526
Title: A Randomized, Controlled, Open-label, Multicenter, Phase IIb Safety and Efficacy Study of rhHNS (Recombinant Human Heparan N Sulfatase) Administration Via an Intrathecal Drug Delivery Device in Pediatric Patients With Early Stage Mucopolysaccharidosis Type IIIA Disease
Brief Title: Randomized, Controlled, Open-label, Multicenter, Safety and Efficacy Study of rhHNS Administration Via an IDDD in Pediatric Patients With Early Stage MPS IIIA Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGT-SAN-093; 2013-003450-24 (EudraCT Number)
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Sanfilippo Syndrome
Keywords: sulfoglucosamine sulfohydrolase (SGSH); recombinant human heparan N-sulfatase (rhHNS); Hunter's Syndrome; Shire HGT; Lysosomal Storage Disease (LSD); Sanfilippo Syndrome Type A (Sanfilippo A); enzyme replacement therapy (ERT)
MeSH Terms: conditions — Mucopolysaccharidosis III; Mucopolysaccharidosis II; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 45 mg Q2W (Active Comparator): rhHNS 45 mg administered intrathecally Q2W (once every 2 weeks ie, every 14 days), for 48 weeks via the surgically implanted IDDD (or LP)
  Interventions: Drug: Recombinant human heparan N-sulfatase [rhHNS]
- 45 mg Q4W (Active Comparator): rhHNS 45 mg administered intrathecally Q4W (once every 4 weeks ie, every 28 days), for 48 weeks via the surgically implanted IDDD (or LP)
  Interventions: Drug: Recombinant human heparan N-sulfatase [rhHNS]
- Placebo (Placebo Comparator): The comparator group will receive no treatment with rhHNS.
  Interventions: Drug: Recombinant human heparan N-sulfatase [rhHNS]

INTERVENTIONS:
Drug: Recombinant human heparan N-sulfatase [rhHNS] — Recombinant human heparan N-sulfatase [rhHNS]

SUMMARY:
Sanfilippo syndrome Type A, or Mucopolysaccharidosis (MPS) IIIA, is a rare lysosomal storage disease caused by deficiency of the enzyme heparan N-sulfatase (sulfamidase). In the absence of this enzyme, there is an accumulation of the glycosaminoglycan, heparan sulfate, resulting in progressive neurodegeneration. Symptoms are usually first noted in the 1st or 2nd year of life, although definitive diagnosis is often delayed, with an average age of diagnosis of 4.5 years. The disease is characterized by developmental delays initially, followed by neurological developmental arrest, then regression. These developmental deficits are typically associated with severe behavioral disturbances. Patients have a significantly reduced lifespan, with few surviving beyond the 2nd or 3rd decade.

The purpose of this study is to evaluate the safety and efficacy of recombinant human heparan-N-sulfatase (rhHNS) in pediatric patients with Early Stage Mucopolysaccharidosis Type III A Disease.

DETAILED DESCRIPTION:
No effective, disease-modifying therapies are currently approved as treatments for this devastating and disabling disease.

Shire Human Genetic Therapies (Shire HGT) is developing an enzyme replacement therapy (ERT) recombinant human heparan-N-sulfatase (rhHNS) for patients with MPS IIIA. rhHNS is being administered into the cerebrospinal fluid (CSF) via an surgically implanted intrathecal drug delivery device (IDDD), because when administered intravenously (IV) it does not cross the blood brain barrier (BBB).

This study will evaluate the effect of 48 weeks of rhHNS treatment on the clinical course of MPS IIIA, using cognitive function as the primary outcome measure. The trial will evaluate 2 dosing regimens of rhHNS administered via an IDDD in comparison with a no treatment control group. Patients will be randomized 1:1:1 to either of the treatment groups or the no treatment group. Treatment will be administered in an open-label manner. The safety and tolerability profile of rhHNS will continue to be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following criteria to be enrolled in this study.

1. Documented MPS IIIA diagnosis
2. Age ≥12 months and ≤48 months
3. The patient has a DQ score ≥60%
4. The patient is medically stable, in the opinion of the Investigator, and able to accommodate the protocol requirements, including travel, assessments, and IDDD surgery, without placing an undue burden on the patient/patient's family
5. The patient's parent(s) or legally authorized representative(s) must have voluntarily signed and dated an Independent Ethics Committee-approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient's parent(s), or legally authorized representative(s). Consent of the patient's parent(s) or legally authorized representative(s) must be obtained prior to the start of any study procedures.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study.

1. The presence of significant non-MPS IIIA related CNS impairment or behavioral disturbances that would confound the scientific integrity or interpretation of study assessments, as determined by the Investigator.
2. The presence of at least one S298P mutation in SGSH, associated with attenuated disease OR there is documentation of the S298P mutation in a sibling affected by MPS IIIA, provided parental consent is obtained to use this information.
3. The presence of relatively attenuated MPS IIIA disease in an older sibling, defined as preservation of any speech beyond the age of 10 years.
4. Visual or hearing impairment sufficient, in the clinical judgment of the investigator, to preclude cooperation with neurodevelopmental testing. Use of hearing aids is permitted.
5. In the opinion of the Investigator, the patient is assessed as having an unacceptably high risk for anesthesia due to airway compromise, drug hypersensitivity, or other conditions (such as neuroleptic malignant syndrome, malignant hyperthermia, or other anesthesia-related concerns).
6. The patient has a history of poorly controlled seizure disorder.
7. The patient is currently receiving psychotropic or other medications, which in the Investigator's opinion would be likely to substantially confound test results.
8. The patient has a history of bleeding disorder or is unable to abstain from medications that, in the opinion of the investigator, place them at risk of bleeding following surgery or LP.
9. The patient participated in a clinical trial of another investigational medicinal product, within the 30 days prior to the study (or within 5 elimination half lives of the investigational product), or is currently enrolled in another study that involves an investigational drug or device. NOTE: Nutritional supplements, including genistein are permitted if they are taken or administered outside the context of a formal investigation.
10. The patient has received a hematopoietic stem cell or bone marrow transplant, or gene therapy.
11. The patient has a condition that is contraindicated as described in the SOPH-A-PORT Mini S-IDDD
12. The patient's parent(s) or patient's legally authorized representative(s) is/are unable to understand the nature, scope, and possible consequences of the study, or do/does not agree to comply with the protocol defined schedule of assessments.
13. The patient is unable to comply with the protocol (eg, has a clinically relevant medical condition making implementation of the protocol difficult, unstable social situation, or otherwise unlikely to complete the study) or is, in the opinion of the Investigator, otherwise unsuited for the study.
14. The patient has any item (braces, tattoos, etc.) which would exclude the patient from being able to undergo MRI according to local Institutional Policy, or the patient has any other situation that would exclude the patient from undergoing any other procedure required in this study.

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2014-02-26 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- United States (3):
  - Los Angeles Biomedical Research, Torrance, California
  - University of Minnesota Department of Pediatrics, Minneapolis, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
- Hospital Universitario Austral A Unidad de Investigacion, Buenos Aires, Argentina
- Chu Bicetre, Le Kremlin-Bicêtre, Paris, France
- Universitätsklinikum Hamburg Eppendorf, Hamburg, Germany
- U.O.S Malattie Metaboliche Rare Clinical Pediatrica, Monza, Italy
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Hospital Vall D'Hebron, Barcelona, Spain
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Wijburg FA, Whitley CB, Muenzer J, Gasperini S, Del Toro M, Muschol N, Cleary M, Sevin C, Shapiro E, Bhargava P, Kerr D, Alexanderian D. Intrathecal heparan-N-sulfatase in patients with Sanfilippo syndrome type A: A phase IIb randomized trial. Mol Genet Metab. 2019 Feb;126(2):121-130. doi: 10.1016/j.ymgme.2018.10.006. Epub 2018 Oct 24. PMID 30528227

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 24 participants were screened, of them 21 participants were enrolled in the study.
Groups:
- No HGT-1410: Participants received no treatment (HGT-1410).
- HGT-1410 45 mg Q2W: Participants received HGT-1410 45 milligram (mg) intrathecally once every two weeks (Q2W) using surgically implanted intrathecal drug delivery device (IDDD) or lumbar puncture (LP) for 48 weeks.
- HGT-1410 45 mg Q4W: Participants received HGT-1410 45 mg intrathecally once every four weeks (Q4W) using surgically implanted IDDD or LP for 48 weeks.
Period: Overall Study
Arm/Group | No HGT-1410 | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Started | 7 | 7 | 7
Completed | 7 | 7 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- HGT-1410 45 mg Q2W: Participants received HGT-1410 45 mg intrathecally Q2W using surgically implanted IDDD or LP for 48 weeks.
- HGT-1410 45 mg Q4W: Participants received HGT-1410 45 mg intrathecally Q4W using surgically implanted IDDD or LP for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | No HGT-1410 | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W | Total
Number analyzed (Participants) | 7 | 7 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: months] | 32.42 (9.548) | 29.64 (9.989) | 33.53 (9.336) | 31.87 (9.287)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 12
  Male | 4 | 2 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response Using Bayley Scales of Infant Development Assessment Third Edition (BSID-III)
Description: The BSID--III is a series of measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers and consists of a series of developmental play tasks. The development quotient (DQ) is a means to express a neurodevelopmental/cognitive delay which was computed as a ratio and expressed as a percentage using the age equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range: 0, 100). The BSID--III DQ score is based on the cognitive domain. A positive value indicates improvement in health and cognition. Overall response was the maximum decline in the DQ of 10 points or less over 48 weeks. Number of participants with the overall response were reported here.
Time Frame: Baseline (Week 0) up to Week 48
Population: ITT population included all randomized participants.
Measure: Number; unit: participants
Arm/Group | No HGT-1410 | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Number analyzed (Participants) | 7 | 7 | 7
participants | 0 | 2 | 1
Statistical Analysis 1: Comparison: No HGT-1410 vs HGT-1410 45 mg Q2W; 95% exact unconditional confidence interval of the difference in proportion between each of the treatment groups and the untreated control group was considered for the parameter estimation; Test type: Superiority or Other; p = 0.4615, Fisher Exact; Difference between proportions = 0.286, 95% CI 2-sided [-0.297 to 0.745]
Statistical Analysis 2: Comparison: No HGT-1410 vs HGT-1410 45 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Difference between proportions = 0.143, 95% CI 2-sided [-0.423 to 0.647]

2. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE)
Description: An adverse event (AE) was any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered investigational product related. This included an exacerbation of a pre-existing condition. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline (Week 0) up to Week 52
Population: Safety population included all participants who received a dose of HGT-1410 either using IDDD implantation or LP; underwent the IDDD surgical implant procedure without receiving a dose of HGT-1410; were randomly assigned to the untreated group and had any safety follow-up data.
Measure: Number; unit: participants
Arm/Group | No HGT-1410 | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Number analyzed (Participants) | 7 | 7 | 7
participants | 3 | 5 | 6

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered investigational product related. This included an exacerbation of a pre-existing condition. TEAEs were defined as AE occurring on or after the time of first IDDD implantation or LP procedure to the end of study (EOS) visit (+30 days).
Time Frame: Baseline (Week 0) up to Week 52
Population: Safety population included all participants who received a dose of HGT-1410 using the IDDD implantation or LP; underwent the IDDD surgical implant procedure without receiving a dose of HGT-1410; were randomly assigned to the untreated group and had any safety follow-up data.
Measure: Number; unit: participants
Arm/Group | No HGT-1410 | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Number analyzed (Participants) | 7 | 7 | 7
participants | 6 | 7 | 7

4. Secondary Outcome: Number of Participants With Positive Anti-recombinant Human Heparan-N-Sulfatase (rhHNS) Antibody in Serum at Week 48
Description: A participant was considered positive if they had at least 1 positive result during the study. Once a participant reported antibody positive, they were considered positive for the remainder of the study.
Time Frame: Baseline (Week 0) up to Week 48
Population: Safety population included all participants who received a dose of HGT-1410 using either the IDDD implantation or LP; underwent the IDDD surgical implant procedure without receiving a dose of HGT-1410; were randomly assigned to the untreated group and had any safety followup data.
Measure: Number; unit: participants
Arm/Group | No HGT-1410 | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Number analyzed (Participants) | 7 | 7 | 7
participants | 1 | 7 | 6

5. Secondary Outcome: Change From Baseline in Vineland Adaptive Behavior Scales Second Edition (VABS-II) Development Quotient (DQ) Score at Week 48
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. The DQ is a means to express a neurodevelopmental/cognitive delay. The DQ was computed as a ratio and expressed as a percentage using the age-equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range, 0, 100). The overall DQ score is calculated from the mean age-equivalent score obtained by averaging out the age-equivalent scores for the all the sub-domains except for Gross and Fine motor skills. This test measures the following 5 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite (a composite of the other 4 domains). A positive value indicates improvement in health and cognition.
Time Frame: Baseline (Week 0), Week 48
Population: ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: percentage of chronological age
Arm/Group | No HGT-1410 | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Number analyzed (Participants) | 7 | 7 | 7
percentage of chronological age
  Communication Domain: number analyzed (Participants) | 7 | 6 | 7
  Communication Domain | -5.12 (10.981) | -20.83 (23.475) | -4.97 (17.253)
  Daily Living Skills Domain: number analyzed (Participants) | 6 | 6 | 6
  Daily Living Skills Domain | -4.20 (29.005) | -27.09 (21.444) | -11.74 (26.713)
  Socialization Domain: number analyzed (Participants) | 6 | 6 | 6
  Socialization Domain | -16.12 (23.320) | -24.24 (40.617) | -29.34 (29.425)
  Motor Skills Domain: number analyzed (Participants) | 6 | 6 | 6
  Motor Skills Domain | -5.37 (24.741) | -27.01 (20.820) | -17.88 (12.007)

6. Secondary Outcome: Change From Baseline in Development Quotient (DQ) Using Bayley Scales of Infant Development Assessment Third Edition (BSID-III) at Week 48
Description: The BSID--III is a series of measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers and consists of a series of developmental play tasks. The DQ is a means to express a neurodevelopmental/cognitive delay which was computed as a ratio and expressed as a percentage using the age-equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range: 0, 100). The BSID--III DQ score is based on the cognitive domain. A positive value indicates improvement in health and cognition.
Time Frame: Baseline (Week 0), Week 48
Population: ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: percentage of chronological age
Arm/Group | No HGT-1410 | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Number analyzed (Participants) | 7 | 7 | 7
percentage of chronological age
  Cognitive | -19.81 (3.974) | -23.82 (14.684) | -19.87 (12.724)
  Receptive Communication | -13.15 (13.318) | -16.33 (25.373) | -12.41 (14.981)
  Expressive Communication | -14.77 (10.055) | -19.71 (22.878) | -10.01 (15.573)
  Fine Motor | -23.72 (14.752) | -18.59 (18.879) | -18.86 (16.308)
  Gross Motor | -11.60 (13.668) | -12.52 (21.203) | -2.77 (18.947)

7. Secondary Outcome: Change From Baseline in Total Cortical Grey Matter Volume at Week 48
Description: The change from baseline in grey matter volume at Week 48 was assessed by magnetic resonance imaging (MRI).
Time Frame: Baseline (Week 0), Week 48
Population: ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: cubic centimeter (cc)
Arm/Group | No HGT-1410 | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Number analyzed (Participants) | 7 | 7 | 7
cubic centimeter (cc) | -45.1 (23.35) | -102.0 (68.12) | -58.8 (66.24)

8. Secondary Outcome: Change From Baseline in Concentration of Glycosaminoglycan (GAG) in Cerebrospinal Fluid (CSF) at Week 48
Description: Change from baseline in concentration of GAG in CSF at Week 48 was reported.
Time Frame: Baseline (Week 0), Week 48
Population: ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | No HGT-1410 | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Number analyzed (Participants) | 7 | 7 | 7
micromolar | -0.193 (1.318) | -6.888 (5.388) | -5.924 (2.470)

9. Secondary Outcome: Change From Baseline in Concentration of GAG in Urine at Week 48
Description: The concentration of GAG in urine was normalized to the urine creatinine value and reported as milligram (mg) GAG per millimole (mmol) creatinine.
Time Frame: Baseline (Week 0), Week 48
Population: ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: mg GAG/mmol creatinine
Arm/Group | No HGT-1410 | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Number analyzed (Participants) | 7 | 7 | 7
mg GAG/mmol creatinine | -7.18 (39.175) | -31.81 (22.887) | -42.46 (29.861)

10. Secondary Outcome: Concentration of Recombinant Human Heparan-N-Sulfatase (rhHNS) in Cerebrospinal Fluid (CSF)
Description: Concentration of rhHNS in CSF was assessed using validated enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Pre-dose, 4, 48 hours on Week 0 and Week 48
Population: Pharmacokinetic (PK) population included all participants who received HGT-1410, participated in the scheduled PK studies, and had sufficient samples available for analysis.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/ml)
Arm/Group | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Number analyzed (Participants) | 7 | 7
nanogram per milliliter (ng/ml)
  Week 0: Predose | 0 (0) | 0 (0)
  Week 0: 4h: number analyzed (Participants) | 5 | 5
  Week 0: 4h | 313392.49 (142748.885) | 266021.60 (113340.887)
  Week 0: 48h: number analyzed (Participants) | 6 | 6
  Week 0: 48h | 366.05 (571.528) | 2119.59 (2068.093)
  Week 48: Predose: number analyzed (Participants) | 6 | 7
  Week 48: Predose | 869.67 (1863.989) | 365.04 (965.797)
  Week 48: 4h: number analyzed (Participants) | 5 | 5
  Week 48: 4h | 374544.38 (135047.700) | 335203.84 (82918.537)
  Week 48: 48h: number analyzed (Participants) | 4 | 5
  Week 48: 48h | 104.49 (65.881) | 8892.93 (19519.717)

11. Secondary Outcome: Maximum Observed Drug Concentration (Cmax) of Recombinant Human Heparan-N-Sulfatase (rhHNS) in Serum
Description: Cmax of rhHNS in serum was evaluated using enzyme-linked immunosorbent assay (ELISA) method and liquid chromatography tandem mass spectrometry (LC-MS) method.
Time Frame: Predose, 0.5 h, 1 h, 2 h, 4 h, 8 h, 12 h, 24 h, and 48 h post-dose on Week 0 and Week 48
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Number analyzed (Participants) | 7 | 7
ng/ml
  ELISA Method: Week 0 | 120.9 (84.77) | 237.0 (159.68)
  ELISA Method: Week 48: number analyzed (Participants) | 7 | 4
  ELISA Method: Week 48 | 63.5 (149.76) | 118.8 (161.98)
  LC-MS Method: Week 0 | 102.4 (63.00) | 191.0 (125.84)
  LC-MS Method: Week 48: number analyzed (Participants) | 7 | 5
  LC-MS Method: Week 48 | 188.1 (127.40) | 119.7 (133.18)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Week 52
Arm/Group | No HGT-1410 | HGT-1410 45 mg Q2W | HGT-1410 45 mg Q4W
Serious Adverse Events (participants affected / at risk) | 3/7 | 5/7 | 6/7
Other Adverse Events (participants affected / at risk) | 6/7 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No HGT-1410 (N=7) | HGT-1410 45 mg Q2W (N=7) | HGT-1410 45 mg Q4W (N=7)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (8) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device breakage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device failure (General disorders) | 0 (0) | 1 (1) | 1 (1)
Implant site extravasation (General disorders) | 0 (0) | 2 (3) | 0 (0)
Implant site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Central nervous system infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Incision site swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No HGT-1410 (N=7) | HGT-1410 45 mg Q2W (N=7) | HGT-1410 45 mg Q4W (N=7)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rickets (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diastolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Diastolic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 5 (12) | 3 (4)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Developmental delay (General disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Implant site extravasation (General disorders) | 0 (0) | 1 (1) | 2 (4)
Implant site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (10) | 4 (22) | 4 (5)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (4) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 2 (3) | 0 (0) | 4 (6)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (3) | 1 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Hand-Foot-And-Mouth disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (6) | 0 (0) | 2 (4)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (4) | 1 (3) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (3) | 3 (4) | 1 (2)
Scarlet fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Stitch abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (6) | 5 (18) | 1 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 1 (1) | 0 (0) | 1 (5)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure systolic decreased (Investigations) | 1 (1) | 0 (0) | 1 (10)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Body temperature decreased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Crystal urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Csf protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Csf test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Csf white blood cell count increased (Investigations) | 0 (0) | 1 (2) | 3 (3)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 1 (1) | 0 (0) | 1 (2)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (8)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 1 (5) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Protein total increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Respiratory rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Urine uric acid (Investigations) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Demyelination (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Drooling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Motor dysfunction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Sleep terror (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mucocutaneous rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.